CLINICAL TRIAL: NCT05013697
Title: A Multicenter Exploratory Study of Paclitaxel+Cisplatin+TQB2450 Injection Combined With or Without Anlotinib in the First-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: TQB2450 Solution for Injection (TQB2450)+Paclitaxel+Cisplatin ± Anlotinib in the Treatment of Esophageal Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-13
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group 1 (Experimental): Initial treatment: Paclitaxel + Cisplatin + TQB2450 injection+ Anlotinib (4-6 cycles).
  Maintenance treatment: TQB2450 injection+Anlotinib.
  Interventions: Drug: Paclitaxel + Cisplatin + TQB2450 injection+ Anlotinib
- Experimental group 2 (Experimental): Initial treatment: Paclitaxel + Cisplatin + TQB2450 injection (4-6 cycles). Maintenance treatment: TQB2450 injection.
  Interventions: Drug: Paclitaxel + Cisplatin + TQB2450 injection

INTERVENTIONS:
Drug: Paclitaxel + Cisplatin + TQB2450 injection+ Anlotinib — TQB2450 injection: 1200 mg, i.v.gtt , d1;Anlotinib 10mg, po.qd , d1-14；Paclitaxel 135mg/m2, i.v.gtt , d1; Cisplatin 60-75mg/m2, i.v.gtt , d1-d3; The above schemes are repeated every three weeks. After 4-6 cycles, the regimen is changed to Anlotinib (10mg, po.qd , d1-14)+TQB2450 injection（1200 mg, i.v.gtt , d1）. The regimen is repeated every 3 weeks until the disease progresses.
  Arms: Experimental group 1
Drug: Paclitaxel + Cisplatin + TQB2450 injection — TQB2450 injection: 1200 mg, i.v.gtt , d1;Paclitaxel 135mg/m2, i.v.gtt , d1; Cisplatin 60-75mg/m2, i.v.gtt , d1-d3; The above schemes are repeated every three weeks. After 4-6 cycles, the regimen is changed to TQB2450 injection（1200 mg, i.v.gtt , d1）. The regimen is repeated every 3 weeks until the disease progresses.
  Arms: Experimental group 2

SUMMARY:
The regimen of paclitaxel+cisplatin+TQB2450 injection combined or not combined with anlotinib is the first-line treatment of advanced esophageal squamous cell carcinoma. Take PFS as the main evaluation index, the purpose is to evaluate its effectiveness and safety

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the esophagus, locally advanced, unresectable, recurrent or metastatic disease.
* Those who have not received systemic treatment before, or who relapsed after (new) adjuvant therapy/radical surgery more than 6 months ; Note: Including advanced or recurrent Patients who ever received only radiotherapy on non-target lesions. The duration from the end of palliative treatment for local lesions (non-target lesions) to enrollment should > 2 weeks;
* According to RECIST 1.1, at least one measurable lesion; the measurable lesions should not have received local treatment such as radiotherapy (for the lesions in the area where received local radiotherapy, it can also be regarded as a target lesion if confirmed to progress according to the recist1.1);
* 18 and 75 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1；Life expectancy of at least 3 months.
* the main organ function to meet the following criteria:

  (1)Blood routine tests met the following requirements:

  a) haemoglobin(HB)≥90g/L ； b) absolute neutrophil count(NEUT)≥1.5×109/L ； c) platelet count(PLT)≥100×109/L；

  （2） Biochemical tests met the following requirements： total bilirubin(TBIL)≤ 1.5 times the upper limit of normal (ULN) .≤5 × ULN if with liver involvement； serum creatinine ≤1.5 × the ULN or creatinine clearance≥50mL/min。

  （3） Coagulation or thyroid function meet the following criteria: International Normalized Ratio (INR) ≤1.5 and Partial Thromboplastin Time (PT) or activated PTT (APTT) ≤1.5 × (ULN))."
* Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study
* The patient volunteers to participate in the study, signs a consent form, has good compliance, and obeys the follow-up, and is willing and able to follow the protocol during the study.

Exclusion Criteria:

* Patients tends to have complete obstruction or patients requiring interventional treatment for obstruction;
* Patients with a high risk of bleeding or perforation due to the apparent invasion of adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed fistulas;
* Patients with symptoms of hematemesis, hematochezia and daily bleeding ≥ 2.5 mL, or any bleeding event with Common Terminology Criteria for Adverse Events （CTCAE） level 3 within 3 months before screening;
* allergic to study drugs 、paclitaxel and cisplatin preparations or excipients;
* Adjuvant chemotherapy patients who have used paclitaxel or cisplatin, and relapse or metastasize within one year
* A variety of factors affecting oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* patients with any severe and / or uncontrolled disease, including:Unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmhg or diastolic blood pressure ≥100) Mmhg) patients; patients with grade ≥ myocardial ischemia or myocardial infarction, arrhythmia (including qt interval ≥ 480ms); according to nyha criteria, iii-iv cardiac dysfunction, or cardiac ultrasonography prompted left ventricular ejection fraction (lvef) <50% of patients;live Severe infection that is sexual or uncontrolled;Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;poor diabetes control (fasting blood glucose (fbg)>10mmol/l);Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g
* long-term unhealed wounds or fractures;
* Patients with active hemorrhage within 2 months of primary lesions; pulmonary hemorrhage with NCI CTCAE grade >1, 4 weeks before of enrollment; other sites of bleeding NCI CTCAE grade >2, 4 weeks before of enrollment; patients with bleeding tendency (such as active gastrointestinal ulcers) or patients undergoing thrombolytic or anticoagulant therapy such as warfarin, heparin or its analogues;
* Have undergone major surgery (craniotomy, thoracotomy or open surgery) within 4 weeks prior to the first dose study or Major surgery is required during the study period.
* A history of gastrointestinal perforation and/or fistula occurred within 6 months prior to treatment; or an overactive/venous thrombosis event such as a cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and lung Embolism；
* Symptomatic central nervous system metastasis and/or cancerous meningitis are known to exist;
* Clinically significant ascites, including any ascites that can be found on a physical examination, ascites that has been treated or currently in need of treatment, and only those with a small amount of ascites but no symptoms can be selected;
* A moderate amount of fluid in both sides of the chest, or a large amount of fluid in one side of the chest, or has caused respiratory dysfunction Patient to be drained;
* known to have active tuberculosis;
* suffering from interstitial lung disease requiring steroid therapy;
* Uncontrolled metabolic disorders or other non-malignant tumors or systemic diseases or cancer secondary reactions that can lead to higher medical risks and/or survival Evaluation of uncertainty;
* Significantly malnourished patients;
* those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* A history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
* History of other primary malignancies, but the following : 1) complete remission of malignant tumors for at least 2 years prior to enrollment and no additional treatment during the study; 2) non-melanoma skin cancer or malignant freckle-like sputum with adequate treatment and no evidence of disease recurrence; 3) adequately treated and In situ carcinoma without evidence of disease recurrence;
* Female patients who are pregnant or breastfeeding;
* According to the judgment of the investigator, there is a concomitant disease that seriously endangers the safety of the patient or affects the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS， RECIST assessment) | each 42 days（Initial treatment） or 63 days ( Maintenance treatment) up to Progressive Disease or Intolerable toxicity （Up to 24 months）

SECONDARY OUTCOMES:
Progression-free survival (iPFS) | each 42 days（Initial treatment） or 63 days ( Maintenance treatment) up to Progressive Disease or Intolerable toxicity （Up to 24 months）
Objective response rate (ORR) | each 42 days（Initial treatment） or 63 days ( Maintenance treatment) up to Progressive Disease or Intolerable toxicity （Up to 24 months）
Disease control rate (DCR） | each 42 days（Initial treatment） or 63 days ( Maintenance treatment) up to Progressive Disease or Intolerable toxicity （Up to 24 months）
Duration of response (DOR) | each 42 days（Initial treatment） or 63 days ( Maintenance treatment) up to Progressive Disease or Intolerable toxicity （Up to 24 months）
Incidence of Treatment-related adverse Events | Through study completion, an average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Doctor, Study Chair — Henan Cancer Hospital
Locations (5):
- China (5):
  - AnYang Tumor Hospital, Anyang, Henan
  - The People's Hospital Of AnYang City, Anyang, Henan
  - First Affiliated Hospital of Henan University of Science and Technolog, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lu D, Ni Z, Liu X, Feng S, Dong X, Shi X, Zhai J, Mai S, Jiang J, Wang Z, Wu H, Cai K. Beyond T Cells: Understanding the Role of PD-1/PD-L1 in Tumor-Associated Macrophages. J Immunol Res. 2019 Nov 4;2019:1919082. doi: 10.1155/2019/1919082. eCollection 2019. PMID 31781673
- [Background] Ramjiawan RR, Griffioen AW, Duda DG. Anti-angiogenesis for cancer revisited: Is there a role for combinations with immunotherapy? Angiogenesis. 2017 May;20(2):185-204. doi: 10.1007/s10456-017-9552-y. Epub 2017 Mar 30. PMID 28361267
- [Background] [1]He Jie, Shao Kang. The epidemiology, diagnosis and treatment of esophageal cancer in China and future strategies[J]. Chinese Journal of Cancer, 2011, 21(07): 501-504.
- [Result] Gandini S, Massi D, Mandala M. PD-L1 expression in cancer patients receiving anti PD-1/PD-L1 antibodies: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2016 Apr;100:88-98. doi: 10.1016/j.critrevonc.2016.02.001. Epub 2016 Feb 10. PMID 26895815
- [Result] Chen W, Sun K, Zheng R, Zeng H, Zhang S, Xia C, Yang Z, Li H, Zou X, He J. Cancer incidence and mortality in China, 2014. Chin J Cancer Res. 2018 Feb;30(1):1-12. doi: 10.21147/j.issn.1000-9604.2018.01.01. PMID 29545714
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Guidelines Working Committee of Chinese Society of Clinical Oncology. Guidelines for Diagnosis and Treatment of Esophageal Cancer (2021 Edition) [M]. Beijing: People's Medical Publishing House, 2021.
- [Result] Blot, W. J. & Tarone, R. E. Esophageal cancer. Nat Rev Dis Prim. 3, 17048 (2017).
- [Derived] Li N, Xia J, Gao X, Zhou J, Hong Y, Cui D, Zhao X, Wu T, Guo Y, Wang J, Luo S. First-line benmelstobart plus anlotinib and chemotherapy in advanced or metastatic/recurrent esophageal squamous cell carcinoma: a multi-center phase 2 study. Signal Transduct Target Ther. 2024 Nov 8;9(1):303. doi: 10.1038/s41392-024-02008-7. PMID 39511164